CLINICAL TRIAL: NCT04795830
Title: Clinical and Radiographic Evaluation of Bioactive Materials in Pulp Therapy of Primary Teeth: A Randomized Controlled Trial
Brief Title: Bioactive Materials in Pulp Therapy of Primary Teeth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Hisham Abdelwahab, Assistant Lecturer of Pediatric Dentistry and Dental Public Health, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED 20-5D
Record Dates: First submitted 2021-02-21; First posted 2021-03-12 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Pulpitis; Pulp Disease, Dental
Keywords: Pulpitis; Pulp Inflammation; Primary dentition; bioceramic; root repair material; deciduous dentition; pulpotomy; MTA; bioactive
MeSH Terms: conditions — Pulpitis; Dental Pulp Diseases | interventions — Pulpotomy; mineral trioxide aggregate

STUDY DESIGN:
Intervention Model Description: After informed consent, baseline clinical and radiographic assessment will be obtained and recorded in the patient's examination sheet. Enrolled participant's tooth will be then randomly allocated to the experiment or control intervention group. Participant will be recalled for follow up assessments at 1, 3, 6 and 12 months. A 14 day window, defined as 7 days before and 7 days after the due date, will be available to complete the 1 and 3 month follow-up evaluations and a 28 day window, defined as 7 days before and 21 days after the due date, will be available to complete the 6 and 12 month follow up evaluations.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to which group they are assigned to. Both materials used have the same white color and any labels on syringes will be hidden with appropriate wrap. Teeth treated will be assigned codes so that outcome evaluators at follow up appointments are blinded. Furthermore, baseline clinical and radiographic findings of sound teeth as well as after pulp therapy and stainless steel crown placement will not reveal the material being used at the intervention, since the stainless steel crown obscures the view clinically and radiographically. On the other hand, the operator/primary investigator cannot be blinded as she is already familiar with the nature of the materials used and their different modes of application. For statistical analysis, codes will also assure blinding and confidentiality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group with Stainless Steel Crown (SSC) (Active Comparator): After pulpotomy and hemostasis, MTA powder and liquid will be mixed according to the manufacturer's instructions and applied via MTA applicator to cover the amputated pulp stumps.
  Using a glass ionomer gun, a capsule of GC Corporation's EQUIA Forte High Translucency glass ionomer restorative (GC EQUIA Forte HT Fil Capsule) will be injected to fill the pulp chamber.
  Finally, the tooth will be restored with a stainless steel crown.
  Interventions: Combination Product: Mineral Trioxide Aggregate as pulp dressing in primary molars (MTA)
- Control group with Restoration (Active Comparator): After pulpotomy and hemostasis, MTA powder and liquid will be mixed according to the manufacturer's instructions and applied via MTA applicator to cover the amputated pulp stumps.
  Using a glass ionomer gun, a capsule of glass ionomer restorative GC EQUIA Forte HT Fil Capsule will be injected to fill the pulp chamber and restore the tooth.
  Interventions: Combination Product: Mineral Trioxide Aggregate as pulp dressing in primary molars (MTA)
- Study group with Restoration (Experimental): After pulpotomy and hemostasis, BC RRM Fast setting putty will be applied from the manufacturer's syringe using a plastic instrument to cover the amputated pulp stumps.
  Using a glass ionomer gun, a capsule of glass ionomer restorative GC EQUIA Forte HT Fil Capsule will be injected to fill the pulp chamber and restore the tooth.
  Interventions: Combination Product: Bioceramic root repair material as pulp dressing in pulpotomy in primary molars
- Study group with Stainless Steel Crown (SSC) (Experimental): After pulpotomy and hemostasis, BC RRM Fast setting putty will be applied from the manufacturer's syringe using a plastic instrument to cover the amputated pulp stumps.
  Using a glass ionomer gun, a capsule of glass ionomer restorative GC EQUIA Forte HT Fil Capsule will be injected to fill the pulp chamber.
  Finally, the tooth will be restored with a stainless steel crown.
  Interventions: Combination Product: Bioceramic root repair material as pulp dressing in pulpotomy in primary molars

INTERVENTIONS:
Combination Product: Bioceramic root repair material as pulp dressing in pulpotomy in primary molars — BC RRM-F, a novel premixed bioceramic-based putty, can be used as a pulp dressing to promote pulp healing and repair with an added convenience for the pediatric patient. The aim of the present study is to evaluate the efficacy of a bioceramic root repair material as pulp dressing in pulpotomy in primary molars. The success of this material as pulpotomy dressing in primary molars will be evaluated clinically and radiographically in comparison to mineral trioxide aggregate pulpotomy. Both materials will be compared in terms of ease of handling, time to perform procedure and convenience of application. Each material's success will be evaluated by comparing its performance with or without the added peripheral seal of a stainless steel crown.
  Other Names: Bioceramic Root Repair Material Fast Set Putty (BC RRM-F); TotalFill® BC RRM™ Fast Set Putty, FKG Dentaire SA, Switzerland
  Arms: Study group with Restoration; Study group with Stainless Steel Crown (SSC)
Combination Product: Mineral Trioxide Aggregate as pulp dressing in primary molars (MTA) — MTA's sealing ability, biocompatibility, ability to stimulate hard tissue formation and its regenerative ability when used in contact with pulp tissues has made MTA pulpotomy the new gold standard as opposed to formocresol pulpotomy in treating the amputated pulp stumps of primary molars.
  Other Names: PD™ MTA WHITE, Produits Dentaires SA, Switzerland
  Arms: Control group with Restoration; Control group with Stainless Steel Crown (SSC)

SUMMARY:
The purpose of this study is to compare the clinical and radiographic success of a new injectable, fast setting bioceramic root repair material (BC RRM) putty with mineral trioxide aggregate (MTA) in pulpotomy procedures of primary teeth. The null hypothesis (H0) is that there is no difference in the clinical and radiographic success between the TotalFill® BC RRM™ Fast Set Putty and Produits Dentaires™ (PD™) MTA WHITE when used as a pulp dressing in pulpotomies of primary molars.

DETAILED DESCRIPTION:
Dental Caries is the most common chronic disease worldwide and the most common disease of childhood, with increasing prevalence in many countries, including Egypt. About 70% of Egyptian children have some untreated caries experience. This percentage was also reported by an unpublished nationwide survey funded by the World Health Organization (WHO).

Dental decay is the primary cause for oral pain and tooth loss. Toothache as a result of untreated caries is persistent and often severe. In children, the prevalence of dental pain ranges from 5% to 33% and increases with caries severity, child age and decreasing economic status. Untreated caries in children can lead to pain, sepsis and affect the quality of life of children and their families, such as lost school days, family disruption, and the need for costly dental treatment.

Tooth decay has a multifactorial nature of occurrence. The carious process is a result of an imbalance between pathogenic factors, namely the high frequency of fermentable sugar intake and the increase in acid-producing bacteria, which outweigh host protective factors in the oral cavity favoring demineralization of the tooth structure. This on-going process progresses more rapidly in primary compared to permanent teeth which may be attributed to the different anatomical characteristics between them. Thinner enamel and dentin as well as larger pulp and higher pulp horns make deciduous teeth more vulnerable to degradation of hard tissues and pulpal affection. Approximately 75% of deep carious lesions were found clinically with pulp exposure.

The deciduous teeth are important for mastication, speech, esthetics as well as for the preservation of arch integrity and space for the permanent successors. Hence, pulp therapy is the appropriate alternative to extraction for pulpally affected primary teeth in most clinical situations. Depending on the extension of the carious process, different pulp treatment modalities are available, pulpotomy being the most common among them with a high success rate of 82.6%. Complete pulpotomy involves the complete removal of the inflamed and/or infected coronal pulp tissue and the application of a medicament to the pulp chamber or radicular pulp remnants allowing healing of the radicular pulp tissue.

For decades, formocresol had been the gold standard material for pulpotomy procedures in primary teeth until mineral trioxide aggregate (MTA) was introduced. According to several systematic reviews and meta-analysis, MTA presents superior performance and higher success rates compared to other materials in pulpotomy of primary teeth. MTA pulpotomy has become a safe and biocompatible treatment alternative with success rates comparable to formocresol pulpotomy.

Although MTA has been recently considered the gold standard material for pulpotomy procedures, some drawbacks such as poor handling and long setting time are challenging when used as pulpotomy dressing in primary teeth of children. Thus, the evaluation of the clinical and radiographic performance of other materials such as a bioceramic root repair material in a convenient injectable form with faster setting time is of paramount importance for the management of dental caries in the pediatric patient.

Evidence is lacking as to the effectiveness of bioceramic materials as pulp dressing in the primary dentition and to their clinical or radiographic success compared to other materials. Different bioceramic root repair materials (BC RRM) have been used in the adult population. To our knowledge, there are no studies evaluating the use of BC RRM in pulp therapy of deciduous molars. Since MTA has been recently advocated to be the gold standard in pulp therapy, it is chosen as the comparator in the control group.

A two arm, parallel group, randomized controlled trial, with 1:1 allocation ratio to either study group or control group, is the study of choice to test the null hypothesis and answer the research question.

The study will be conducted at the outpatient clinic of the department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Ain Shams University. This research will be reviewed by the Research Ethics Committee and Institutional Review Board, Faculty of Dentistry, Ain Shams University. A verbal as well as a written consent will be obtained from the caregivers of the participants after explaining the objectives of the study and assuring complete confidentiality of data. All caregivers and participants will be informed that they have the right to withdraw from the study at any time. Moreover, participants 6 years and older will be requested to sign an assent form after an age appropriate explanation of the trial procedures and their objectives. All consent and assent forms are translated into Arabic.

A power analysis was designed to have adequate power to apply a statistical test of the research hypothesis (null hypothesis) that there was no difference between the clinical and radiographic success between the bioceramic root repair material and Mineral Trioxide Aggregate when used as a pulp dressing in pulpotomies of primary molars. By adopting an alpha (α) level of 0.05 (5%), a beta (β) level of 0.20 (20%) i.e. power=80%, and using an effect size (w=0.430); the predicted sample size (n) was found to be a total of (52) teeth; i.e. (26) for each group and (13) for each subgroup. Sample size calculation was performed using G*Power version 3.1.9.2.44 The sample size was increased by 15% to (30) primary molars per group, i.e. (15) molars per subgroup and (60) in total to compensate for drop-outs.

The study interventions are expected to be conducted from 2020 until 2022. After informed consent, baseline clinical and radiographic assessment will be obtained and recorded in the patient's examination sheet. Enrolled participant's tooth will be then randomly allocated to the experiment or control intervention group. Participant will be recalled for follow up assessments at 1, 3, 6 and 12 months. A 14 day window, defined as 7 days before and 7 days after the due date, will be available to complete the 1 and 3 month follow-up evaluations and a 28 day window, defined as 7 days before and 21 days after the due date, will be available to complete the 6 and 12 month follow up evaluations.

Participants' data will be recorded in an examination sheet and stored as hard copy files. Patients' information will be regarded as confidential and will never be revealed at all times. This will be ensured by assigning codes to participants' teeth undergoing intervention.

Several attempts will be made calling participants on the phone for clinical and radiographic follow up appointments at 1, 3, 6 and 12 months. Patients who fail to show up at the follow up examinations, within the defined follow up windows, will be automatically excluded from the study. Patients who are no longer willing to continue in the study have the right to quit at any time and will be offered to continue dental treatment at the department's outpatient clinic.

All data will be collected, tabulated, summarized and statistically analyzed using the Statistical Packages for Social Sciences (SPSS) software.

Regular unannounced audits by the Research Ethics Committee, Faculty of Dentistry, Ain Shams University are expected as to ascertain that protocol guidelines are followed throughout the study. In addition to the study supervisors, independent staff members and clinic supervisors of the Department of Pediatric Dentistry and Dental Public Health, Ain Shams University monitor clinical performance to ensure adherence to best practice.

MTA and BC RRM have been shown to have no adverse effects on healthy patients. On the contrary, they have been shown to be biomimetic and biocompatible when used for endodontic procedures in adults. Failure of pulp therapy and abscess formation might occur as with all materials used in pulpotomies to this date. Short term follow up will avoid the occurrence of any serious condition and will allow its instant treatment. Any adverse event will be recorded and managed promptly. Furthermore, in case of consistent failures, the use of the experimental material will be stopped and patients will be treated with another modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a restorable vital deep carious primary molar which is indicated for pulpotomy
* Absence of clinical signs and symptoms; namely pain on percussion, tooth mobility, presence of sinus or fistula or history of swelling

Exclusion Criteria:

* Badly broken down, unrestorable teeth
* Teeth with previous pulp therapy treatment
* Presence of uncontrolled bleeding
* Clinical evidence of non-vitality; namely presence of an abscess or a sinus tract or premature mobility
* Radiographic evidence of bone resorption, internal or external root resorption, or periapical or interradicular radiolucency.
* Uncooperative patients

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical Success of Pulpotomy Treatment after 1 month follow up | 1 month
  During the follow-up phase, clinical outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  1-month evaluation
  Clinical findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following clinical findings indicate the success of the material used in pulp therapy. Presence of any of the clinical findings will be considered as a failure of the material used in pulp therapy.
  Clinical findings:
  Pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around crown margins denoting poor oral hygiene Pain on percussion on clinical examination Non-physiologic mobility
Clinical Success of Pulpotomy Treatment after 3 months follow up | 3 months
  During the follow-up phase, clinical outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  3-months evaluation Clinical findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following clinical findings indicate the success of the material used in pulp therapy. Presence of any of the clinical findings will be considered as a failure of the material used in pulp therapy.
  Clinical findings:
  Pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around crown margins denoting poor oral hygiene Pain on percussion on clinical examination Non-physiologic mobility
Clinical Success of Pulpotomy Treatment after 6 months follow up | 6 months
  During the follow-up phase, clinical outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  6-months evaluation Clinical findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following clinical findings indicate the success of the material used in pulp therapy. Presence of any of the clinical findings will be considered as a failure of the material used in pulp therapy.
  Clinical findings:
  Pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around crown margins denoting poor oral hygiene Pain on percussion on clinical examination Non-physiologic mobility
Clinical Success of Pulpotomy Treatment after 12 months follow up | 12 months
  During the follow-up phase, clinical outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  12-months evaluation Clinical findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following clinical findings indicate the success of the material used in pulp therapy. Presence of any of the clinical findings will be considered as a failure of the material used in pulp therapy.
  Clinical findings:
  Pain on mastication or spontaneous pain, as reported by the patient, without clinical evidence of plaque retention around crown margins denoting poor oral hygiene Pain on percussion on clinical examination Non-physiologic mobility
Radiographic Success of Pulpotomy Treatment after 1 month follow up | 1 month
  During the follow-up phase, radiographic outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  1-month evaluation
  Radiographic findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following radiographic findings indicate the success of the material used in pulp therapy. Presence of any of the radiographic findings will be considered as a failure of the material used in pulp therapy.
  Radiographic findings:
  Pathological internal or external root resorption Interradicular or periapical bone loss Interradicular or periapical radiolucency
Radiographic Success of Pulpotomy Treatment after 3 months follow up | 3 months
  During the follow-up phase, radiographic outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  3-months evaluation
  Radiographic findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following radiographic findings indicate the success of the material used in pulp therapy. Presence of any of the radiographic findings will be considered as a failure of the material used in pulp therapy.
  Radiographic findings:
  Pathological internal or external root resorption Interradicular or periapical bone loss Interradicular or periapical radiolucency
Radiographic Success of Pulpotomy Treatment after 6 months follow up | 6 months
  During the follow-up phase, radiographic outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  6-months evaluation
  Radiographic findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following radiographic findings indicate the success of the material used in pulp therapy. Presence of any of the radiographic findings will be considered as a failure of the material used in pulp therapy.
  Radiographic findings:
  Pathological internal or external root resorption Interradicular or periapical bone loss Interradicular or periapical radiolucency
Radiographic Success of Pulpotomy Treatment after 12 months follow up | 12 months
  During the follow-up phase, radiographic outcomes will be evaluated by the primary investigator and two other blinded calibrated examiners at the following timing:
  12-months evaluation
  Radiographic findings will be discussed until all three examiners come to a conclusion of whether the pulp therapy of the tooth was a success or a failure. The absence of the following radiographic findings indicate the success of the material used in pulp therapy. Presence of any of the radiographic findings will be considered as a failure of the material used in pulp therapy.
  Radiographic findings:
  Pathological internal or external root resorption Interradicular or periapical bone loss Interradicular or periapical radiolucency

SECONDARY OUTCOMES:
Ease of handling of material | during procedure
  Both materials will be compared in terms of ease of handling by answering the following Yes or No questions:
  Does the material stick to the plastic instrument when inserted into the cavity? Does the material set before adequate amount is applied to cover pulp stumps (adequate working time)?
Time to perform procedure | during procedure
  Both materials will be compared in terms of time to perform procedure by measuring the time (in minutes) taken to perform the procedure using a stopwatch.
Convenience of application | during procedure
  Both materials will be compared in terms of convenience of application by answering the following Yes or No questions:
  Does the material adapt poorly to the cavity walls when observed by the naked eye? Does the patient feel pain or discomfort when the material is being applied to the pulp stumps?

CONTACTS AND LOCATIONS:
Overall Officials: Dina Abdelwahab, M.Sc., Principal Investigator — Department of Pediatric Dentistry and Dental Public Health, Ain Shams University
Locations (1):
- Outpatient Clinic of the Department of Pediatric Dentistry, Ain Shams University, Cairo, Egypt

REFERENCES:
- [Derived] Abdelwahab DH, Kabil NS, Badran AS, Darwish D, Abd El Geleel OM. One-year radiographic and clinical performance of bioactive materials in primary molar pulpotomy: A randomized controlled trial. J Dent. 2024 Apr;143:104864. doi: 10.1016/j.jdent.2024.104864. Epub 2024 Jan 26. PMID 38281619